CLINICAL TRIAL: NCT03215095
Title: Radioiodine (RAI) in Combination With Durvalumab (Medi4736) for RAI-avid, Recurrent/Metastatic Thyroid Cancers
Brief Title: RAI Plus Immunotherapy for Recurrent/Metastatic Thyroid Cancers
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-218
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Cancer
Keywords: Radioiodine (RAI); Durvalumab (Medi4736); RAI-avid; 17-218
MeSH Terms: conditions — Thyroid Neoplasms | interventions — durvalumab; Iodine-131

STUDY DESIGN:
Intervention Model Description: This is a pilot study with the primary objective to assess the safety of administering the PD-L1 targeting agent durvalumab in combination with recombinant human thyroid stimulating hormone (rhTSH, Thyrogen) stimulated/prepared radioiodine (RAI; 131I) therapy in patients with RAI-avid (RAIA) recurrent and/or metastatic (R/M) thyroid cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radioiodine (RAI) in Combination with Durvalumab (Medi4736) (Experimental): Enrolled patients will be treated with durvalumab 1500 mg IV every 4 weeks. In Cycle 1/Week 3, Thyrogen 0.9 mg IM will be administered on two consecutive calendar days followed by 100 mCi (+/- 10 mCi) of RAI the next calendar day. Durvalumab will be continued every 4 weeks.
  Interventions: Drug: Durvalumab (Medi4736); Radiation: Radioiodine (RAI)

INTERVENTIONS:
Drug: Durvalumab (Medi4736) — durvalumab 1500 mg IV every 4 weeks
Radiation: Radioiodine (RAI) — 100 mCi (+/- 10 mCi) of 131I will be administered a day after Thyrogen injections have been administered for two consecutive calendar days.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, a drug called durvalumab combined with Thyrogen-stimulated RAI, has on the patient and thyroid cancer. Durvalumab is a drug that has been developed to activate the immune system by blocking a protein called programmed death ligand-1 (PD-L1) that can be present on tumor and normal cells, including immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed thyroid carcinoma of follicular origin (including papillary, follicular, hurthle cell or poorly differentiated subtypes and their respective variants).
* Diagnosis of recurrent and/or metastatic thyroid cancer
* At least one RAI-avid lesion identified on the most recent radioiodine scan (a diagnostic, post-therapy, or post-ablation scan) OR at least one lesion on the most recent FDG PET scan with an SUV max of 10 or less. (Both RAI-sensitive and RAI-refractory patients are eligible if at least one tumor with RAI avidity of any degree can be identified within one of these parameters.)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease. Tumors in previously irradiated fields may be considered measureable if there is evidence of tumor progression after radiation treatment.
* ECOG Performance Status (PS) 0 or 1. (or Karnofsky ≥60%)
* Age ≥ 18 years at time of study entry
* Adequate normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
  * Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). (This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
  * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
* Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) . 72 x serum creatinine (mg/dL)

* Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patients must agree to undergo two research biopsies of (a) malignant lesion(s). Biopsies do not need to be done if the investigator or person performing the biopsy judges there is no tumor accessible for biopsy, the only accessible tumor must be used for RECIST measurement, or the biopsy poses too great a risk to the patient. If the patient has only one RECIST measureable target lesion for response assessment, research biopsies must not be performed on that target lesion.
* Availability of archival tumor tissue from the thyroid cancer primary or metastasis (a tissue block or a minimum of 30 unstained slides would be required. Patients with less archival tissue available may still be eligible for the study after discussion with the MSK Principal Investigator.)

Exclusion Criteria:

* 131I therapy < 6 months prior to initiation of therapy on this protocol. A diagnostic study using < 10 mCi of 131I is not considered 131I therapy.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
* History of pneumonitis.
* External beam radiation therapy < 4 weeks prior to initiation of therapy on this protocol.
* Chemotherapy, immunotherapy, targeted therapy, monoclonal antibodies, tumor embolization, or other investigational agent within 28 days prior to the first dose of study drug.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity CTCAE grade ≥ 2 from previous anti-cancer therapy. Exceptions include hearing loss, peripheral neuropathy, and alopecia.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with a history of autoimmune thyroid disease are not excluded. Subjects with vitiligo or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to durvalumab or any excipient.
* History of hypersensitivity to thyrotropin alpha (Thyrogen).
* Patients unable to follow a low iodine diet or requiring medication with high content in iodide (amiodarone).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known history of active tuberculosis.
* Symptomatic brain metasteses, leptomeningeal carcinomatosis, or spinal cord compression (treated metastatic brain, leptomeningeal carcinomatosis, or spinal cord compression are allowed). Note: Patients must be off steroids used for brain metasteses, leptomeningeal carcinomatosis, or spinal cord compression.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radioiodine (RAI) in Combination With Durvalumab (Medi4736)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radioiodine (RAI) in Combination With Durvalumab (Medi4736)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 67 [53 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-Limiting Toxicity (DLTs)
Description: Grading of DLTs will follow the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 6 weeks beginning from the first durvalumab
Measure: Count of Participants; unit: Participants
Arm/Group | Radioiodine (RAI) in Combination With Durvalumab (Medi4736)
Number analyzed (Participants) | 11
Participants
  Participants with DLTs | 0
  Participants with no DLTs | 11

2. Secondary Outcome: Best Overall Response
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radioiodine (RAI) in Combination With Durvalumab (Medi4736)
Number analyzed (Participants) | 11
Participants
  Partial Response | 2
  Stable Disease | 7
  Progressive Disease | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Radioiodine (RAI) in Combination With Durvalumab (Medi4736)
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radioiodine (RAI) in Combination With Durvalumab (Medi4736) (N=11)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Weight loss (Investigations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Paresthesia (Nervous system disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Neutrophil Count Decrease (Investigations) | 1
Fatigue (General disorders) | 3
Hypertension (Vascular disorders) | 1
Platelet Count Decrease (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03215095/Prot_SAP_000.pdf